CLINICAL TRIAL: NCT06695702
Title: The Effect of Collaborative Learning Approach with Concept Maps on Nursing Students' Knowledge Learning on Symptom Management in Cancer Patients: a Randomized Controlled Study
Brief Title: Cancer Symptom Management in Nursing Students
Status: Completed | Type: Observational
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Other Study IDs: Aysun Acun 11
Record Dates: First submitted 2024-11-14; First posted 2024-11-19 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-11

CONDITIONS: Nursing Students
Keywords: oncology; nursing student; Collaborative Learning Approach
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- nursing students' level of knowledge about oncology symptoms: The benefit of workbased learning on nursing students' knowledge of oncology symptom management
  Interventions: Other: the effect of work-based learning on the level of knowledge

INTERVENTIONS:
Other: the effect of work-based learning on the level of knowledge — The benefit of workbased learning on nursing students' knowledge of oncology symptom management

SUMMARY:
Ensuring that nursing students learn the symptoms seen in cancer.

DETAILED DESCRIPTION:
Nursing education plays an important role in providing the knowledge, skills and critical thinking abilities needed to provide quality care. Innovative teaching strategies provide quality education. These methods, such as cooperative learning and concept maps, help them to criticize and apply their knowledge. It is important to integrate these strategies in oncology nursing education, which involves complex treatment processes and symptom management. Collaborative learning with concept maps can contribute to the development of a more holistic understanding of oncology care. This study was planned to examine the effect of collaborative learning approach with concept maps on nursing students' knowledge learning about symptom management of oncologic patients.

ELIGIBILITY:
Inclusion Criteria:

* The sample of the study will consist of students who were attending the course on the date the research data were collected,
* who had not received education for oncology patients before and
* who agreed to participate in the study.
* It will be aimed to include all students who meet the inclusion criteria.

Exclusion Criteria:

* Students who were absent from the course and
* did not participate in the pre-test, post-test and follow-up test will be excluded from the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: nursing students
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
questionnaire on knowledge of oncologic symptoms | 14/11/2024-31/12/2024
  nursing students' level of knowledge

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)